CLINICAL TRIAL: NCT01736501
Title: Surveying Parents About Genome Screening of Newborns
Acronym: BabySeq
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This was not a clinical trial.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Robert C. Green, MD, MPH, Lecturer on Medicine & Associate Director for Research, Partners Center for Personalized Genetic Medicine, Brigham and Women's Hospital
Allocation: Randomized | Masking: None
Other Study IDs: 2012-P-001197
Record Dates: First submitted 2012-11-01; First posted 2012-11-29 (Estimated); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Parents of Healthy Newborns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Baseline1-demographics (No Intervention): Baseline survey- demographics only
- Baseline1 w/genetics (Other): Genetics education, baseline interest in genome screening - 1
  Interventions: Other: Genetics education at baseline
- Baseline2-demographics (Other): Baseline survey- demographics only
  Interventions: Other: Hypothetical genomic scenarios at follow-up
- Baseline2 w/genetics (Other): Genetics education, baseline interest in genome screening - 2
  Interventions: Other: Genetics education at baseline; Other: Hypothetical genomic scenarios at follow-up

INTERVENTIONS:
Other: Genetics education at baseline
  Arms: Baseline1 w/genetics; Baseline2 w/genetics
Other: Hypothetical genomic scenarios at follow-up
  Arms: Baseline2 w/genetics; Baseline2-demographics

SUMMARY:
A 10 minute baseline survey will be administered to parents of healthy newborn infants while in the hospital after delivery at Brigham and Women's Hospital, to be followed by a 25 minute survey 3-24 months later. We will measure parents' attitudes and preferences related to genome screening of newborns. The specific aims of this study are:

1. To investigate whether parents' opinions regarding genome screening of newborns change between the first 48 hours post-partum and 3-24 months post-partum.

   a. We hypothesize that there will not be significant differences between interest in genome screening results in the 48 hours post-partum compared to 3-24 months post-partum.
2. To determine whether seeing hypothetical genome screening results affects parents' decisions regarding whether they would want genome screening for their newborn.

   1. We expect many parents to state initially (in the 48 hours post-partum) that they would elect to have genome screening for their newborn if it were available. In the follow-up survey, half of study participants will receive hypothetical scenarios in which they will need to struggle with the probabilistic and ambiguous nature of the information that could be derived from genome sequencing. We will examine whether this alters their preferences. We will also explore whether parents who receive hypothetical genome screening results scenarios are more likely to alter their preferences than parents who do not receive hypothetical scenarios.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a healthy newborn in the BWH Department of Obstetrics
* English-speaking

Exclusion Criteria:

* Impaired decision-making capacity
* Newborn with life-threatening health concerns in the 48 hours post-partum

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Interest in genome screening for newborn if this service were available through a research study | Change between baseline and 3-24 month follow-up
  This is a question created by the investigators. It uses a 5-point Likert scale to measure parents' self-reported interest in genome screening for their newborn.

SECONDARY OUTCOMES:
Rate of refusal of newborn screening | baseline
  Newborn screening refusals are very rare. When they occur, they are tracked by nurses on the postpartum inpatient unit. At the start of all shifts for study recruitment, the research assistant will ask the nurse-in-charge if any patients refused newborn screening since the previous study recruitment shift.

OTHER OUTCOMES:
Parental Stress | 3-28 month follow-up
  Parenting Stress Index- short form
Postpartum bonding | 3-28 month follow-up
  Postpartum Bonding Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Green, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Waisbren SE, Back DK, Liu C, Kalia SS, Ringer SA, Holm IA, Green RC. Parents are interested in newborn genomic testing during the early postpartum period. Genet Med. 2015 Jun;17(6):501-4. doi: 10.1038/gim.2014.139. Epub 2014 Dec 4. PMID 25474344